CLINICAL TRIAL: NCT02889042
Title: Repeated Voluntary Drug Intoxication (IMVr): Characterization of a New Addictive Behavior by Clinical Phenotyping and Functional Imaging
Acronym: Phenot IMVr
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC14.182
Record Dates: First submitted 2016-08-03; First posted 2016-09-05 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Volunteers Repeated Drug Poisoning; Alcoholic; Volunteers
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Volunteers repeated drug poisoning (Experimental): performing MRI and a biological assessment
  Interventions: Other: MRI and biological assessment
- Volunteers single drug poisoning (Other): performing MRI and a biological assessment
  Interventions: Other: MRI and biological assessment
- alcoholic (Other): performing MRI and a biological assessment
  Interventions: Other: MRI and biological assessment
- volunteers (Other): performing MRI and a biological assessment
  Interventions: Other: MRI and biological assessment

INTERVENTIONS:
Other: MRI and biological assessment — performing a MRI and a biological assessment

SUMMARY:
France is one of the European countries with the highest rate of death by suicide, more than 10 400 deaths each year, about 16 people out of 100 000. Although suicide mortality rate tends to fall between 1987 and 2008 the number of suicide attempts (TS) against observed by an upward trend between 2005 and 2010. However, the most important predictor of death by suicide remains the TS. Now these are primarily TS Poisoning Drug-Volunteer (IMV), especially benzodiazepines. These IMV, there have been 16% recurrence in the past year and 21% at 4 years among hospitalized patients. Or a Health Barometer 2005 survey showed that 58% of respondents with a TS over the last 12 months had not been hospitalized. This type of acting out, especially the repeated IMV (IMVr) is underestimated epidemiologically because it is an unknown phenomenon and too little screened by health professionals.

DETAILED DESCRIPTION:
The IMVr constitute severe behavior disorder, chronic and costly given the multiple prescriptions, hospital admissions, including emergencies, and repeated treatment failures, in the absence of specific treatment of psychopathological problematic background. Indeed many arguments lead to evoke the existence of a functioning underlying addictive type, rather than a problem of suicide, especially from the second recurrence (often characterized by low lethality and suicidal intentionality). This impulsive behavior and / or compulsive repeatedly would not simply the consequence of a pharmacological benzodiazepine dependence (it is also not systematic), but would demonstrate a similar operation to that of behavioral addictions. Furthermore, a preliminary study has shown that this type of behavior was not limited to a BPD personality type, since it is mainly found pathological personalities depressive and avoidant types.

In this context it is urgent to make an accurate characterization of these patients IMVr because the integration of the addictive dimension in their care will adapt strategies psychotherapeutic, pharmacological, and the terms of issue of psychotropic and especially benzodiazepines .

ELIGIBILITY:
Inclusion Criteria:

Will be offered for study subjects that meet the following criteria:

* Man or woman hospitalized (e) in the aftermath of a IMV:

  * History of at least 2 for the IMV group IMVr
  * First suicide attempt high intentionality (SIS score> 20/30) for group IMVS
* Man or woman with alcohol dependence according to DSM-IV-TR, in the aftermath of withdrawal (outpatient or inpatient) for the alcohol group
* Man or woman free from any addictive disorder, suicidal or mood for the control group

And all of the following criteria:

* Age greater than or equal to 18 and less than or equal to 60 years
* Informed consent in writing signed by the patient
* Person affiliated to the social security or beneficiary of such a scheme

Exclusion Criteria:

For IMVS Group:

* Have a history of scarification or addictive disorder (behavioral or product)

In the alcohol group:

* TS present history

For all patients, presenting at least one of the following criteria:

* Age less than 18 years, over 60 years.
* acute or chronic delusional disorder.
* Cognitive impairment or impeding the reading comprehension quizzes.
* secondary pathologies at a stroke.
* Denial of participation.
* Contraindications to MRI.
* Subjects with clinically significant gastrointestinal, renal, hepatic, endocrine, cardiovascular or respiratory (especially persistent asthma) which can prevent stay of 60 min in MRI without being hindered.
* No participant to another pharmacological study.
* unauthorized treatments: all psychotropic treatments (except anti-anxiety treatments benzodiazepine average duration of action and antihistamine), baclofen and other treatment can modify vasoreactivity fMRI.
* Coagulation disorders against-indicating blood.
* People under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Comparison of local measurements of changes in the BOLD (Blood Oxygenation Level Dependent) based on visual stimuli by anatomical and functional MRI | 15 days of the passage to the act

CONTACTS AND LOCATIONS:
Overall Officials: PENNEL Lucie, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided